CLINICAL TRIAL: NCT01547884
Title: Effect of Filarial Infection on Antigen-Specific Immune Responses in Latent Tuberculosis
Brief Title: Effect of Filarial Infection on Immune Responses in Latent Tuberculosis
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999912073; 12-I-N073
Record Dates: First submitted 2012-03-06; First posted 2012-03-08 (Estimated); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Mycobacterium Infections; Tuberculosis; Filariasis; Latent Tuberculosis
Keywords: T Cells; Immune Responses; Mycobacterial Antigens; Tissue-invasive Helminth Parasites; Cytokines
MeSH Terms: conditions — Mycobacterium Infections; Tuberculosis; Filariasis; Latent Tuberculosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Latent TB positive with helminth positive
- 2: Latent TB positive with helminth negative

SUMMARY:
Background:

- Lymphatic filariasis is an infection that is caused by small, thread-like worms. It is spread by mosquitoes, and causes fever, chills, and headaches. If untreated, it can also cause elephantiasis, a condition that leads to swelling of the arms, legs, breasts, and scrotum. Treatment can eliminate the worms from the blood and reduce the risk of developing elephantiasis. Researchers want to study people with latent tuberculosis (TB) who may or may not be infected with filariasis. This study will look at the way that people with latent TB fight infection with these worms.

Objectives:

- To study how the immune systems of people with latent TB react to filarial infection.

Eligibility:

- Individuals between 18 and 65 years of age who have latent TB and may or may not have filarial infection.

Design:

* Participants will be screened with a physical exam and medical history. They will provide a blood and stool sample to test for infection.
* Participants who do not have lymphatic filariasis but have another kind of intestinal worm will be treated for the parasite. This will be their last study visit.
* Participants who have latent TB and lymphatic filariasis will be treated with the standard treatment for the disease. They will come back for a second visit 6 months later, and will provide another blood sample.

DETAILED DESCRIPTION:
Tissue-invasive helminth parasites infect close to 500 million people worldwide and are associated with strong T helper (Th)2 responses and regulatory networks that downregulate potentially protective Th1 responses. The two common tissue invasive helminth parasites are Wuchereria bancrofti, that causes lymphatic filariasis and Strongyloides stercoralis, that causes stronyloidiasis. Previous studies have shown that the intestinal helminth coinfection is accompanied by lowered in vitro production of interferon-gamma and elevated production of interleukin 10 in individuals with active pulmonary tuberculosis (TB). Our team has recently shown that co-existent filarial TB infections down-regulate Th1 and Th17 responses, which are necessary for protection against active TB.

The current study will compare immune responses to mycobacterial antigens in individuals with latent tuberculosis (LTBI+) and concomitant helminth infection (Hel+), including those with filarial (Fil+) and strongyloides (STR+) infection versus those with LTBI+ without concomitant helminth infection (Hel-). Immune responses to mycobacterial antigens from co-infected individuals will also be evaluated before and after treatment for helminth infection. Individuals (n=4000) will sign a screening consent prior to undergoing any study procedures. Every participant will have their medical history collected and will undergo a physical exam and a tuberculin 2TU purified protein derivative (PPD) skin test; women of childbearing potential will also undergo a urine pregnancy test, and those with positive test results will be excluded from the study. Individuals with positive PPD skin test results (> or = 5 mm) and no symptoms of active TB will have their blood drawn (5 mL) as part of the screening procedures to confirm LTBI+ status, evaluate circulating filarial antigenemia, determine Strongyloides status by ELISA, measure hematocrit levels, and for storage of serum samples; those with PPD skin test results less than or equal to 5 mm will be excluded from the study. Individuals with positive symptoms for TB will also be excluded from the study, but sputum will be collected from them, and those with positive smears will be referred for treatment. Individuals will be matched for age, gender, and geographic location, and they will be assigned to one of two groups, LTBI+ Hel+ (n=100) or LTBI+ Hel- (n=100).

Within 3 months of screening, individuals will be asked to sign an on-study consent and will undergo a second blood draw (10 mL) for immunological investigations and storage of serum samples; women of childbearing potential will undergo a repeat urine pregnancy test, and those with positive test results will be excluded from further study. Stool samples will also be collected for microscopic evaluation of ova and parasites. LTBI+ Fil+ individuals will be treated with a single standard dose of albendazole (400 mg) and single standard dose of diethylcarbamazine citrate (300 mg), which are available through the National Programme for the Elimination of Lymphatic Filariasis in India. LTBI+ STR+ individuals will be treated with a single standard dose of ivermectin (12mg) and a single standard dose of albendazole (400mg). These individuals will be asked to return 6 months after treatment to undergo a third blood draw (10 mL) for additional immunological investigations and storage of serum samples. LTBI+ Hel-individuals who test positive for other intestinal helminth infection will be treated with a single standard dose of albendazole (400 mg).

ELIGIBILITY:
* PARTICIPANT INCLUSION CRITERIA:

Individuals (18 to 65 years of age) who meet the following criteria are eligible to participate in the study:

* Positive tuberculin PPD skin test result (>or equal to 5 mm) and IGRA+.
* Willingness to provide blood and stool samples for examination.
* Willingness to have samples stored for study participants only.

PARTICIPANT EXCLUSION CRITERIA:

Individuals are not eligible to participate if:

* Pulmonary symptoms suggestive of TB (cough >3 weeks in duration and/or intermittent fever >1 week in duration and/or hemoptysis).
* Tuberculin skin test within the last 6 months prior to screening.
* Women who are pregnant or breastfeeding.
* Known documented cases of cancer, acquired immune deficiency syndrome, or other immunosuppressive illness.
* History of any other illness or condition which, in the investigator s judgment, may substantially increase the risk associated with the subject s participation in the protocol, or it may compromise the scientific objectives.
* Consumption of DEC in the last one year prior to screening.
* EXCLUSION OF PREGNANT WOMEN:
* Pregnancy: Pregnant and lactating women will be excluded from the study because the safety of DEC or ivermectin has not been adequately evaluated during pregnancy or lactation, while albendazole is a Category C drug found to be teratogenic in animals, and it poses a potential risk during breastfeeding.
* EXCLUSION OF CHILDREN: Children (<18 years of age) will not be included in this study due to the fact the prevalence of filarial and strongyloides infection in children has been found to be very low in South India.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The screening will be a community-based study in South India. Study participants will be recruited from villages in the Kancheepuram District, where approximately 6% of the population tests positive for circulating filarial antigens [31]. PPD skin test reactivity in this population is virtually 100% to PPD-B (battery) and 60% to 70% to PPD-S (standard) by age 24, and the incidence of active TB is about 4 per 1000 individuals [31]. While the rate of positivity of the tuberculin skin test to the 2TU PPD test is not known, significant deviation in the percent positivity from skin tests using 1TU is not expected based on findings reported elsewhere [32]. However, we are revising the @@@screening sample number on the basis of preliminary data from the current study that shows that the prevalence of latent TB in this population is around 25% and filariasis is around 1%. In addition, preliminary data from these areas show that the prevalence of Stronglyloides infection is around 10%.
Sampling Method: Non-Probability Sample
Enrollment: 4268 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2020-08-07 (Actual)

PRIMARY OUTCOMES:
To compare the immune responses to mycobacterial antigens, including PPD and Mycobacterium tuberculosis culture filtrate protein, in individuals who are LTBI+ Hel- versus those who are LTBI+Hel+ | 5 years
  pending

SECONDARY OUTCOMES:
To compare immune responses to mycobacterial antigens in LTBI+ Hel+ co- infected individuals, before and after treatment for filarialinfection. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Thomas B Nutman, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (2):
- National Institute of Allergy and Infectious Diseases (NIAID), 9000 Rockville Pi, Bethesda, Maryland, United States
- Nih-Nirt Icer, Chennai, India

REFERENCES:
- [Background] Metenou S, Babu S, Nutman TB. Impact of filarial infections on coincident intracellular pathogens: Mycobacterium tuberculosis and Plasmodium falciparum. Curr Opin HIV AIDS. 2012 May;7(3):231-8. doi: 10.1097/COH.0b013e3283522c3d. PMID 22418448
- [Background] Babu S, Nutman TB. Helminth-Tuberculosis Co-infection: An Immunologic Perspective. Trends Immunol. 2016 Sep;37(9):597-607. doi: 10.1016/j.it.2016.07.005. Epub 2016 Aug 5. PMID 27501916
- [Background] Salgame P, Yap GS, Gause WC. Effect of helminth-induced immunity on infections with microbial pathogens. Nat Immunol. 2013 Nov;14(11):1118-1126. doi: 10.1038/ni.2736. PMID 24145791